CLINICAL TRIAL: NCT05099991
Title: Transcervical Balloon Compared to Osmotic Dilators Prior to Surgical Abortion: a Non-Inferiority Randomized Trial
Brief Title: Transcervical Balloon Compared to Osmotic Dilators Prior to Surgical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-63172
Record Dates: First submitted 2021-10-17; First posted 2021-10-29 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Abortion, Second Trimester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dilapan-S (Placebo Comparator): A number of Dilapan-S will be inserted for cervical preparation. The number will be determined by a standard protocol that is based on gestational age. The dilators will stay in until the next day prior to their procedure, or earlier if they fall out on their own.
  Interventions: Device: Dilapan-S
- Foley balloon (Experimental): A Foley balloon will be inserted for cervical preparation and filled to 30mL of water or saline. The balloon will stay in until the next day prior to their procedure, or earlier if it falls out on its own.
  Interventions: Device: Single Foley Balloon

INTERVENTIONS:
Device: Single Foley Balloon — Foley Balloon will be placed through the cervix and inflated with 30mL of saline or water on the day prior to the procedure
  Arms: Foley balloon
Device: Dilapan-S — Dilapan S will be placed through the cervix on the day prior to the procedure
  Arms: Dilapan-S

SUMMARY:
The purpose of this study is to determine whether a Foley balloon is similar to osmotic dilators for preparing the cervix prior to a second trimester abortion. Procedure time will be used to compare the two different methods of cervical preparation, reflecting the ease at which the surgeon can perform through a prepared cervix. The aim is to expand effective options for cervical preparation that will can accommodate for varying patient characteristics and provider experiences.

ELIGIBILITY:
Inclusion Criteria:

* presenting to clinic for second trimester abortion at 18 to 23 weeks and 6 days gestation confirmed by ultrasound
* able to provide informed consent and comply with study protocol
* English or Spanish-speaking
* candidate for outpatient cervical preparation

Exclusion Criteria:

* Anyone with an allergy to misoprostol, mifepristone or any study medication
* premature rupture of membranes
* intrauterine fetal demise
* placenta previa
* suspected abnormal placentation
* evidence of infection at the time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu SM, Henkel A, Meza P, Shorter JM, Cahill E, Blumenthal PD, Shaw KA. Comparing transcervical balloon with osmotic dilators for cervical preparation prior to procedural abortion: A noninferiority randomized trial. Contraception. 2024 Dec;140:110550. doi: 10.1016/j.contraception.2024.110550. Epub 2024 Jul 25. PMID 39067560

RESULTS

PARTICIPANT FLOW:
Groups:
- Dilapan-S: Dilapan-S for cervical preparation, number determined by a standard protocol based on gestational age.
- Foley Balloon: Foley balloon inserted for cervical preparation and filled to 30mL of water or saline.
Period: Overall Study
Arm/Group | Dilapan-S | Foley Balloon
Started | 16 | 16
Received Allocated Intervention | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dilapan-S | Foley Balloon | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (3.9) | 32.7 (7.0) | 34.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could select more than one option to indicate they identify with more than one race, ethnicity, or nationality.
  Participants
    American Indian/Alaska Native | 1 | 0 | 1
    White | 6 | 5 | 11
    Black or African American | 1 | 2 | 3
    Asian or Indian | 5 | 0 | 5
    Chinese | 0 | 1 | 1
    Japanese | 0 | 1 | 1
    Korean | 0 | 1 | 1
    Vietnamese | 1 | 0 | 1
    Mexican | 2 | 5 | 7
    Other Hispanic/Latin Origin | 1 | 1 | 2
    Other Pacific Islander | 0 | 1 | 1
    Other | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time
Description: Time to speculum in to speculum out
Time Frame: Up to approximately 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dilapan-S | Foley Balloon
Number analyzed (Participants) | 16 | 16
minutes | 22.4 (12.8) | 22.6 (8.9)
Statistical Analysis 1: Comparison: Dilapan-S vs Foley Balloon; Test type: Non-Inferiority — Non-inferiority would be demonstrated with a mean increase in procedure of 5 minutes; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-7.8 to 8.2]

2. Secondary Outcome: Cervical Dilation
Description: Measure the cervical dilation after removal of the Foley balloon or Dilapan-S
Time Frame: Beginning of the procedure (approximately 5 seconds to assess)
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan-S | Foley Balloon
Number analyzed (Participants) | 16 | 16
Participants
  <1 cm | 0 | 2
  1 cm | 0 | 4
  2 cm | 4 | 3
  3 cm | 6 | 2
  ≥ 4 cm | 6 | 5
Statistical Analysis 1: Comparison: Dilapan-S vs Foley Balloon; Test type: Other; p = 0.07, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 48 hours
Arm/Group | Dilapan-S | Foley Balloon
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dilapan-S (N=16) | Foley Balloon (N=16)
Hemorrhage from atony (Injury, poisoning and procedural complications) | 0 | 1
Cervical abrasion (Injury, poisoning and procedural complications) | 2 | 1
Cervical laceration (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT05099991/Prot_SAP_000.pdf